CLINICAL TRIAL: NCT05999331
Title: Elevated Initial APRI Value Was Associated With the Development of Sepsis-associated Liver Dysfunction in Adult Patients With Sepsis
Brief Title: Elevated Initial APRI Value Was Associated With SALD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Other Study IDs: 2023-06-03
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-06

CONDITIONS: Liver Dysfunction; Sepsis-associated Liver Dysfunction
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-SALD group: SALD did not occur in adult patients with sepsis during ICU stay.SALD was diagnosed by the following criteria: (1) ALT or AST≥20 folds upper limit of normal level; or (2) TBIL≥2.0 mg/dL.
  Interventions: Other: initial aspartate aminotransferase (AST) to platelet (PLT) ratio index
- SALD group: SALD was occured in adult patients with sepsis during ICU stay.SALD was diagnosed by the following criteria: (1) ALT or AST≥20 folds upper limit of normal level; or (2) TBIL≥2.0 mg/dL. SALD is further divided into hypoxic hepatitis and sepsis induced cholestasis (SIC), based on the presence or absence of elevated TBIL. Hypoxic hepatitis is diagnosed when elevated transaminase (>800 IU/L) is present only; and SIC is diagnosed when TBIL is elevated (≥2.0 mg/dL).
  Interventions: Other: initial aspartate aminotransferase (AST) to platelet (PLT) ratio index

INTERVENTIONS:
Other: initial aspartate aminotransferase (AST) to platelet (PLT) ratio index — All eligible patients were given antibiotics therapy, actively control infection source, as well as other supportive therapy to maintain organ function.

SUMMARY:
Sepsis, characterized by severe organ dysfunction related to a dysregulated immune response to infection, is often life-threatening in clinical settings. Sepsis can progress to multiple organ dysfunction syndrome (MODS), causing a great risk of mortality. As a vital immune and metabolic organ, liver often suffers damage in this process and often associated with severe adverse consequences. Compared to general sepsis population, sepsis-associated liver dysfunction (SALD) has a higher mortality, up to 68.6%.

The aspartate aminotransferase (AST) to platelet (PLT) ratio index (APRI), which can be calculated from conventional laboratory indicators, has long been used in the evaluation of liver damage and fibrosis in patients with hepatitis and nonalcoholic fatty liver disease. AST is a sensitive indicator of early liver function impairment. Additionally, PLT also plays a crucial role in sepsis-induced MODS through regulating inflammation, maintaining tissue integrity, and defending against infection. Study found that APRI was a good predictor of SALD occurrence in pediatric patients with sepsis. Furthermore, APRI has also been used to predict the prognostic in septic patients with no history of chronic liver disease.

We conducted a retrospective study based on data from the Medical Information Mart for Intensive Care IV version 2.2 (MIMIC-IV, v2.2) and our own hospital to explore the potential association of APRI with the occurrence of SALD in adult patients with sepsis. Furthermore, we also evaluated the performance of APRI in hypoxic hepatitis and sepsis induced cholestasis (SIC), which are two subtypes of SALD.

DETAILED DESCRIPTION:
We included adult sepsis patients (≥18 years) as study participants, but only those who had data available for their first hospitalization and first ICU admission were enrolled in our study, if they had multiple admission records in the database. Exclusion criteria include: 1) all types of chronic liver disease; 2) viral hepatitis; 3) primary acute cholangiopathies; 4) cholecystitis; 5) hepatic infarction; 6) liver necrosis; 7) liver trauma; 8) length of ICU stay < 24 hours. Patients without simultaneous AST and PLT data in the first 24 hours after ICU admission were also excluded.

The following indicators were extracted directly or derived from the database(MIMIC IV): age; weight; gender; comorbidity, including hypertension, old myocardial infarct, chronic heart failure, cerebrovascular disease, chronic pulmonary disease, chronic renal disease and diabetes; infection site, including blood, lung, skin and soft tissue, abdominal cavity and urinary tract; disease severity scores within the first day of ICU admission, including Acute Physiology Score III (APS III), Sequential Organ Failure Assessment (SOFA), Logistic Organ Dysfunction Score (LODS), Oxford Acute Severity of illness Score (OASIS) and Simplified Acute Physiology Score II (SAPS II); mean vital signs in first 24h, including heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), respiratory rate (RR), temperature and pulse oxygen saturation (SPO2); treatment received within the first day of ICU admission, including invasive ventilation, vasopressor therapy, renal replacement therapy and parenteral nutrition (PN) support; initial laboratory parameters, including white blood cell (WBC) count, hemoglobin, hematocrit, mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), mean corpuscular volume (MCV), red blood cell (RBC), red blood cell distribution width (RDW), platelet, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TBIL), alkaline phosphatase (ALP), albumin, blood urea nitrogen (BUN), creatinine, bicarbonate, anionic gap, sodium, potassium, chloride, total calcium, glucose, prothrombin time (PT), partial prothrombine time (APTT), international normalized ratio (INR) and APRI; clinical outcome measures, including intensive care unit (ICU) length of stay (LOS), hospital LOS, ICU mortality, in-hospital mortality, and 30-day mortality.

The disease severity scores, including APS III, SOFA, LODS, OASIS, SAPS II, are calculated using the SQL code provided by Johnson et al. APRI is calculated by (AST(IU/L)/ upper limits of normal)/PLT(k/uL)×100. Sepsis is diagnosed according to the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). Briefly, patients with confirmed or suspected foci of infectious and a concurrent SOFA≥2. SALD was diagnosed by the following criteria: (1) ALT or AST≥20 folds upper limit of normal level; or (2) TBIL≥2.0 mg/dL. SALD is further divided into hypoxic hepatitis and sepsis induced cholestasis (SIC), based on the presence or absence of elevated TBIL. Hypoxic hepatitis is diagnosed when elevated transaminase (>800 IU/L) is present only; and SIC is diagnosed when TBIL is elevated (≥2.0 mg/dL). Following the exclusion of ineligible patients, the data underwent a thorough examination, and extreme and erroneous values that failed logical checks were removed. Variables with missing data exceeding 30% of the sample size were excluded. For the remaining variables with missing values, the mean imputation method was applied to address them.

We first used the MIMIC IV database to assess the correlation between APRI and the occurrence of SALD using association analysis. We then validated these results using our own data.

ELIGIBILITY:
Inclusion Criteria:

* adult sepsis patients (≥18 years)

Exclusion Criteria:

* all types of chronic liver disease;
* viral hepatitis;
* primary acute cholangiopathies;
* cholecystitis;
* hepatic infarction;
* liver necrosis;
* liver trauma;
* length of ICU stay < 24 hours;
* Patients without simultaneous AST and PLT data in the first 24 hours after ICU admission.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Briefly, patients with confirmed or suspected foci of infectious and a concurrent SOFA≥2 were diagnosed with sepsis. SALD was diagnosed by the following criteria: (1) ALT or AST≥20 folds upper limit of normal level; or (2) TBIL≥2.0 mg/dL.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of SALD | 30 days after ICU admission
  Whether SALD occurs

SECONDARY OUTCOMES:
mortality | 30 days after ICU admission
  Death at 30 days after ICU

CONTACTS AND LOCATIONS:
Overall Officials: Wenkui Yu, professor, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Institute of General Surgery of Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
The research is not over yet

REFERENCES:
- [Background] Dou J, Zhou Y, Cui Y, Chen M, Wang C, Zhang Y. AST-to-Platelet Ratio Index as Potential Early-Warning Biomarker for Sepsis-Associated Liver Injury in Children: A Database Study. Front Pediatr. 2019 Aug 21;7:331. doi: 10.3389/fped.2019.00331. eCollection 2019. PMID 31497584
- [Background] Zhu X, Hu X, Qin X, Pan J, Zhou W. An elevated Fibrosis-4 score is associated with poor clinical outcomes in patients with sepsis: an observational cohort study. Pol Arch Intern Med. 2020 Dec 22;130(12):1064-1073. doi: 10.20452/pamw.15699. Epub 2020 Dec 4. PMID 33274619